CLINICAL TRIAL: NCT00468754
Title: A Study Comparing Continuous Subcutaneous Insulin Infusion With Multiple Daily Injections With Insulin Lispro and Glargine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RD000275; RD000000275
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2010-06

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (2):
- A (Experimental)
  Interventions: Device: Insulin pumps
- B (Experimental)
  Interventions: Device: Insulin pumps

INTERVENTIONS:
Device: Insulin pumps

SUMMARY:
This trial will compare the metabolic control in type 1 diabetes obtained by continuous infusion of insulin lispro with that obtained by multiple daily injections of insulin lispro and glargine, a long-acting insulin analogue. Patients will be switched to the alternative treatment after 4 months. Glucose variability in the last month of each treatment will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic patients, 18-60 years of age
* Diabetic for >2 years
* Treated with CSII for >=6 months
* HbA1c <8.5%

Exclusion Criteria:

* Treatment with daily insulin injections
* Inability to handle pump therapy
* Untreated retinopathy

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2003-07; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Variability of blood glucose characterised by the standard deviation of the mean blood glucose | Length of study

SECONDARY OUTCOMES:
HbA1c | Length of study
Mean BG during the last month of the respective treatment period | Length of study
Frequency of severe hypoglycemia | Length of study
Daily insulin requirement | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Buhr, Study Director — Disetronic Medical Systems AG
Locations (4):
- Italy (4):
  - Bergamo
  - Brescia
  - Padua
  - Pisa